CLINICAL TRIAL: NCT04592510
Title: Impact of COVID-19 on Pediatric Dental Practice During First, Second And Third Wave Among a Group of Pediatric Dentists : A Cross -Sectional Study
Brief Title: Impact of COVID-19 on Pediatric Dental Practice During First, Second And Third Wave.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Essam El-Deen Abdel Rahim, Principal Investigator, Cairo University
Other Study IDs: y66cyyg6
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV2
Keywords: COVID-19; pediatric dentistry
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of impact of covid-19 on pediatric dental practice during first, second and third wave among a group of pediatric dentists.

DETAILED DESCRIPTION:
On the 11th of March, 2020, COVID-19 (SARS-CoV-2) was declared as a pandemic by the World Health Organization. SARS-CoV-2 is an unpredictable virus that is rapidly transmitting from one country to another, and unfortunately as of today, there is no effective medication or vaccine for the disease control. This virus has gone on to cause one of the most rapidly expanding pandemics with over 9 million people being infected worldwide including the pediatric population.

Due to the unique nature of dentistry, most dental procedures generate significant amounts of droplets and aerosols, posing potential risks of infection transmission. Recent studies have demonstrated the role of the oral mucosa in COVID-19 infection, in addition to expressing the ACE2 receptor in salivary glands in the asymptomatic process in infected saliva, thus being one of the main sources of viruses.

Clinical features of COVID-19 in children include fever and cough, but a large proportion of infected children appears to be asymptomatic and may contribute significantly to transmission. Therefore, it can be assumed that, at this stage in the pandemic, all children and their parents/carers are potentially infective with the potential of cross-infection to dental stuff, parents and the public. This has, in theory, an impact on medical and dental procedures that are Aerosol Generating Procedures.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian pediatric dentists with at least Master's degree.
* Work place located in Egypt.

Exclusion Criteria:

* Participants who refuse to participate.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian pediatric dentists regardless of their place of work, in either private clinics or educational hospitals.
Sampling Method: Probability Sample
Enrollment: 345 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Attitude of pediatric dentists toward treating patients in time of COVID-19. | 6 months
  Measuring device by Questionnaire (Ahmadi, Ebrahimi & Ghorbani, 2020) and (Sinjari et al., 2020). The primary outcome is measured using 5-point likert scale scoring to evaluate pediatric dentists' attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Adel El Bardissy, Study Director — Faculty of Oral and dental medicine, Cairo university; Shaimaa Sabry, Study Chair — Faculty of Oral and dental medicine, Cairo university
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Ahmadi H, Ebrahimi A, Ghorbani F. The impact of COVID-19 pandemic on dental practice in Iran: a questionnaire-based report. BMC Oral Health. 2020 Dec 3;20(1):354. doi: 10.1186/s12903-020-01341-x. PMID 33272261
- [Background] Al-Halabi M, Salami A, Alnuaimi E, Kowash M, Hussein I. Assessment of paediatric dental guidelines and caries management alternatives in the post COVID-19 period. A critical review and clinical recommendations. Eur Arch Paediatr Dent. 2020 Oct;21(5):543-556. doi: 10.1007/s40368-020-00547-5. Epub 2020 Jun 16. PMID 32557183
- [Background] BaniHani A, Gardener C, Raggio DP, Santamaria RM, Albadri S. Could COVID-19 change the way we manage caries in primary teeth? Current implications on Paediatric Dentistry. Int J Paediatr Dent. 2020 Sep;30(5):523-525. doi: 10.1111/ipd.12690. No abstract available. PMID 32722881
- [Background] Cook TM. Personal protective equipment during the coronavirus disease (COVID) 2019 pandemic - a narrative review. Anaesthesia. 2020 Jul;75(7):920-927. doi: 10.1111/anae.15071. Epub 2020 Apr 28. PMID 32246849
- [Background] Dong Y, Mo X, Hu Y, Qi X, Jiang F, Jiang Z, Tong S. Epidemiology of COVID-19 Among Children in China. Pediatrics. 2020 Jun;145(6):e20200702. doi: 10.1542/peds.2020-0702. Epub 2020 Mar 16. PMID 32179660
- [Background] Frauenfelder C, Butler C, Hartley B, Cochrane L, Jephson C, Nash R, Hewitt R, Albert D, Wyatt M, Hall A. Practical insights for paediatric otolaryngology surgical cases and performing microlaryngobronchoscopy during the COVID-19 pandemic. Int J Pediatr Otorhinolaryngol. 2020 Jul;134:110030. doi: 10.1016/j.ijporl.2020.110030. Epub 2020 Mar 30. PMID 32278168
- [Background] Qiu H, Wu J, Hong L, Luo Y, Song Q, Chen D. Clinical and epidemiological features of 36 children with coronavirus disease 2019 (COVID-19) in Zhejiang, China: an observational cohort study. Lancet Infect Dis. 2020 Jun;20(6):689-696. doi: 10.1016/S1473-3099(20)30198-5. Epub 2020 Mar 25. PMID 32220650
- [Background] Sinjari B, Rexhepi I, Santilli M, D Addazio G, Chiacchiaretta P, Di Carlo P, Caputi S. The Impact of COVID-19 Related Lockdown on Dental Practice in Central Italy-Outcomes of A Survey. Int J Environ Res Public Health. 2020 Aug 10;17(16):5780. doi: 10.3390/ijerph17165780. PMID 32785056
- [Background] Sundaram M, Ravikumar N, Bansal A, Nallasamy K, Basavaraja GV, Lodha R, Gupta D, Odena MP, Ashwath RNR, Jayashree M; Intensive Care Chapter of Indian Academy of Pediatrics. Novel Coronavirus 2019 (2019-nCoV) Infection: Part II - Respiratory Support in the Pediatric Intensive Care Unit in Resource-limited Settings. Indian Pediatr. 2020 Apr 15;57(4):335-342. doi: 10.1007/s13312-020-1786-x. Epub 2020 Mar 29. PMID 32238613
- [Background] Xu J, Li Y, Gan F, Du Y, Yao Y. Salivary Glands: Potential Reservoirs for COVID-19 Asymptomatic Infection. J Dent Res. 2020 Jul;99(8):989. doi: 10.1177/0022034520918518. Epub 2020 Apr 9. No abstract available. PMID 32271653
- See also: Royal college of surgeons England 2020. Recommendations for paediatric dentistry during COVID-19 pandemic. — https://www.rcseng.ac.uk/-/media/fles/rcs/fds/guidelines/paediatric-dentistry-covid19.pdf.